CLINICAL TRIAL: NCT03199040
Title: A Randomized Phase 1 Trial of Neoantigen DNA Vaccine Alone vs. Neoantigen DNA Vaccine Plus Durvalumab in Triple Negative Breast Cancer Patients Following Standard of Care Therapy
Brief Title: Neoantigen DNA Vaccine Alone vs. Neoantigen DNA Vaccine Plus Durvalumab in Triple Negative Breast Cancer Patients Following Standard of Care Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Drugs/equipment unavailable and insufficient funding
Sponsor: Washington University School of Medicine (Other)
Collaborators: MedImmune LLC (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201710109; 1R01CA240983-01 (NIH)
Record Dates: First submitted 2017-06-22; First posted 2017-06-26 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-04

CONDITIONS: Triple Negative Breast Cancer; Triple Negative Breast Neoplasms; TNBC - Triple-Negative Breast Cancer; Triple-negative Breast Carcinoma
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoantigen DNA vaccine + Durvalumab (Experimental): * The first neoantigen DNA vaccine injection will take place following the completion of standard of care therapy. The day of the first vaccine injection will be referred to as Day 1
  * The schedule of vaccination is Day 1, Day 29 ± 7, Day 57 ± 7, Day 85 ± 7, Day 113 ± 7, and Day 141 ± 7 with at least 21 days between injection days
  * For patients who are randomized to the neoantigen DNA vaccine plus durvalumab arm, the neoantigen-specific T cell response will be assessed prior to Day 85. If a neoantigen-specific T cell response is present, durvalumab will be started on Day 85, and will be administered Q4W at a dose of 1500 mg over the course of 60 minutes. If a neoantigen-specific T cell response is not present, these patients will be replaced but may continue to receive the neoantigen DNA vaccine on study. They will not be transferred to the vaccine-only arm.
  Interventions: Drug: Durvalumab; Biological: Neoantigen DNA vaccine; Device: TDS-IM system (Inchor Medical Systems); Procedure: Peripheral blood draw
- Neoantigen DNA vaccine (Experimental): * The first neoantigen DNA vaccine injection will take place following the completion of standard of care therapy. The day of the first vaccine injection will be referred to as Day 1
  * The schedule of vaccination is Day 1, Day 29 ± 7, Day 57 ± 7, Day 85 ± 7, Day 113 ± 7, and Day 141 ± 7 with at least 21 days between injection days
  Interventions: Biological: Neoantigen DNA vaccine; Device: TDS-IM system (Inchor Medical Systems); Procedure: Peripheral blood draw

INTERVENTIONS:
Drug: Durvalumab — -Human monoclonal antibody
  Other Names: Imfinzi
  Arms: Neoantigen DNA vaccine + Durvalumab
Biological: Neoantigen DNA vaccine — -The vaccine will be given by the TDS-IM system
Device: TDS-IM system (Inchor Medical Systems) — -At each vaccination time point, patients will receive two injections at separate sites.
  Other Names: Integrated electroporation administration system
Procedure: Peripheral blood draw — -Baseline, following completion of standard of care therapy, Day 1, Day 57, Day 113, Day 159, and 1 year after initiation of neoantigen DNA vaccine therapy

SUMMARY:
This is a single institution, open-label randomized phase 1 trial of neoantigen DNA vaccine alone vs. neoantigen DNA vaccine plus durvalumab in triple negative breast cancer (TNBC) patients following standard of care therapy. Patients with newly diagnosed clinical stage II-III TNBC are eligible for enrollment. Patients will receive standard of care therapy including chemotherapy, surgery and radiation therapy as clinically indicated. Following standard of care therapy, patients will be randomized to receive either a neoantigen DNA vaccine alone, or a neoantigen DNA vaccine + durvalumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of invasive breast cancer.
* ER and PR less than Allred score of 3 or less than 1% positive staining cells in the invasive component of the tumor. Patients not meeting this pathology criteria, but have been clinically treated as having TNBC, may be enrolled at treating physician's discretion.
* HER2 negative by FISH or IHC staining 0 or 1+.
* Consented for genome sequencing
* Clinical stage T1c-T4c, any N, M0 primary tumor by AJCC 7th edition clinical staging prior to neoadjuvant chemotherapy, with residual invasive breast cancer after neoadjuvant therapy.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≥1.
* Adequate organ and marrow function no more than 14 days prior to registration as defined below:

  * absolute neutrophil count ≥1,500/μL
  * platelets ≥100,000/μL
  * hemoglobin ≥ 9.0 g/dL
  * total bilirubin ≤ 1.5 X institutional upper limit of normal
  * AST/ALT ≤2.5 X institutional upper limit of normal
  * serum creatinine clearance >40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
* Body weight > 30 kg.
* Evidence of post-menopausal status or negative urine or serum pregnancy test for female pre-menopausal subjects. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, had chemotherapy-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Able to understand and willing to sign an IRB-approved written informed consent document.

Exclusion Criteria:

* Received chemotherapy, radiotherapy (to more than 30% of the bone marrow or with a wide field of radiation), or biologic therapy within the last 30 days.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Receiving any other investigational agent(s) or has received an investigational agent within the last 30 days.
* Receipt of live attenuated vaccination within 6 months prior to study entry or within 30 days of receiving durvalumab.
* Major surgical procedure within 28 days prior to the first dose of durvalumab. Local surgery of isolated lesions for palliative intent is acceptable.
* Current use or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal, inhaled, and intra-articular corticosteroids or systemic corticosteroids at physiological doses which are not to exceed 10 mg/day of prednisone or an equivalent corticosteroid.
* Known metastatic disease.
* Invasive cancer in the contralateral breast.
* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* History of hypersensitivity to durvalumab or any excipient.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 ms calculated from 3 electrocardiograms (ECGs) (within 15 minutes at 5 minutes apart).
* Any unresolved toxicity NCI CTCAE grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria. Subjects with grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician. Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study physician.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, evidence of any acute or chronic viral illness or disease, or psychiatric illness/social situation that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Subjects with vitiligo or alopecia
  * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Subjects without active disease in the last 5 years may be included but only after consultation with the study physician
  * Subjects with celiac disease controlled by diet alone
* History of pneumonitis or interstitial lung disease.
* History of active primary immunodeficiency.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Subjects with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody (anti-HBc) and absence of HBsAg) are eligible. Subjects positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* History of allogeneic organ transplantation.
* Pregnant or breastfeeding. A negative serum pregnancy test is required no more than 7 days before study entry.
* Subjects of reproductive potential who are not willing to employ effective birth control from screening to 1 year after the last dose of durvalumab.
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥ 5 years before the first dose of study treatment and low potential for risk of recurrence
  * Adequately treated non-melanoma skin cancer of lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis.
* Patient must have no active major medical or psychosocial problems that could be complicated by study participation.
* Subjects with a strong likelihood of non-adherence such as difficulties in adhering to follow-up schedule due to geographic distance from the Siteman Cancer Center should not knowingly be registered.
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for eligible injection sites (left and right medial deltoid region) exceeds 40 mm.
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art.
* Therapeutic or traumatic metal implant in the skin or muscle of either deltoid region.
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, or hepatic or renal functional abnormality as determined by the investigator based on medical history, physical examination, EKG, and/or laboratory screening test
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child, or chronic seizure disorder which is well controlled by medication with no seizures within the last 2 years
* Syncopal episode within 12 months of screening
* Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-11-21 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gillanders, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoantigen DNA Vaccine + Durvalumab | Neoantigen DNA Vaccine
Started | 9 | 9
Completed | 5 | 7
Not Completed | 4 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Only completed 5 out of 6 vaccines | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neoantigen DNA Vaccine + Durvalumab | Neoantigen DNA Vaccine | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Median (Full Range); unit: years] | 54 [35 to 75] | 58 [38 to 66] | 54.5 [35 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Safety of Neoantigen DNA Vaccines Given Alone or in Combination With Durvalumab as Measured by Number of Adverse Events Experienced by Patient
Description: * Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v4.03.
  * Assessment of the safety of neoantigen DNA vaccines will include both clinical observation and laboratory evaluation. Safety will be closely monitored after injection with eight or more clinical and laboratory assessments in the first 24 weeks of the trial
Time Frame: 90 days after completion of treatment (approximately day 259)
Measure: Count of Participants; unit: Participants
Arm/Group | Neoantigen DNA Vaccine + Durvalumab | Neoantigen DNA Vaccine
Number analyzed (Participants) | 9 | 9
Participants
  Grade 1-2 anemia | 3 | 1
  Grade 1-2 chest pain-cardiac | 0 | 1
  Grade 1-2 palpitations | 1 | 0
  Grade 1-2 hypothyroidism | 1 | 0
  Grade 1-2 visual migraine | 0 | 1
  Grade 1-2 abdominal cramps | 1 | 0
  Grade 1-2 constipation | 0 | 1
  Grade 1-2 diarrhea | 0 | 1
  Grade 1-2 dyspepsia | 1 | 0
  Grade 1-2 gastritis | 1 | 0
  Grade 1-2 nausea | 2 | 3
  Grade 1-2 vomiting | 1 | 2
  Grade 1-2 ankle edema | 0 | 1
  Grade 1-2 chills | 2 | 2
  Grade 1-2 edema limbs | 1 | 1
  Grade 1-2 fatigue | 3 | 2
  Grade 1-2 fever | 1 | 2
  Grade 1-2 flu-like symptoms | 1 | 2
  Grade 1-2 injection site pain | 9 | 9
  Grade 1-2 localized edema | 2 | 1
  Grade 1-2 neck edema | 1 | 0
  Grade 1-2 COVID-19 infection | 1 | 0
  Grade 1-2 infection from cat bite | 1 | 0
  Grade 1-2 oral herpes lesions | 0 | 1
  Grade 1-2 port infection | 0 | 1
  Grade 1-2 upper respiratory infection | 2 | 0
  Grade 1-2 urinary tract infection | 1 | 0
  Grade 1-2 wound infection | 1 | 0
  Grade 1-2 broken foot | 0 | 1
  Grade 1-2 bruising | 1 | 0
  Grade 1-2 fall | 1 | 0
  Grade 1-2 spinal fracture | 1 | 0
  Grade 3-5 vascular access complication | 0 | 1
  Grade 1-2 alanine aminotransferase increased | 1 | 1
  Grade 1-2 lymphocyte count decreased | 1 | 2
  Grade 3-5 lymphocyte count decreased | 0 | 1
  Grade 1-2 neutrophil count decreased | 0 | 2
  Grade 1-2 weight gain | 0 | 1
  Grade 1-2 weight loss | 1 | 0
  Grade 1-2 white blood cell decreased | 0 | 2
  Grade 1-2 anorexia | 0 | 1
  Grade 1-2 hyperglycemia | 0 | 1
  Grade 1-2 hyperkalemia | 1 | 0
  Grade 1-2 hypokalemia | 0 | 1
  Grade 1-2 hyponatremia | 1 | 1
  Grade 1-2 arthralgia | 1 | 0
  Grade 1-2 bone pain | 0 | 1
  Grade 1-2 myalgia | 7 | 7
  Grade 1-2 neck pain | 2 | 0
  Grade 1-2 pain in extremity | 1 | 1
  Grade 1-2 dizziness | 3 | 0
  Grade 1-2 headache | 1 | 2
  Grade 1-2 neuralgia | 0 | 1
  Grade 1-2 peripheral sensory neuropathy | 2 | 1
  Grade 1-2 insomnia | 1 | 0
  Grade 1-2 breast pain | 1 | 0
  Grade 1-2 vaginal dryness | 0 | 1
  Grade 1-2 allergic rhinitis | 0 | 1
  Grade 1-2 chest congestion | 1 | 0
  Grade 1-2 cough | 1 | 1
  Grade 1-2 dyspnea | 1 | 0
  Grade 1-2 rhinorrhea | 0 | 1
  Grade 1-2 sore throat | 1 | 0
  Grade 1-2 blanching of fingers on left hand | 0 | 1
  Grade 1-2 candidal rash | 1 | 0
  Grade 1-2 eczema | 0 | 1
  Grade 1-2 nail changes | 0 | 1
  Grade 1-2 nodule on breast | 0 | 1
  Grade 1-2 rash maculo-papular | 0 | 1
  Grade 1-2 skin hyperpigmentation | 0 | 1
  Grade 1-2 bilateral breast fat grafting | 1 | 0
  Grade 1-2 hypertension | 2 | 3
  Grade 1-2 lymphedema | 1 | 0

2. Secondary Outcome: Immune Response to Neoantigen DNA Vaccines Given Alone or in Combination With Durvalumab as Measured by Luminex Assay
Description: -Peripheral blood will be collected at multiple time points before and after vaccination
Time Frame: Up to 1 year after completion of treatment (approximately 1 year and 141 days)
Population: The luminex assay was not able to be performed.
Arm/Group | Neoantigen DNA Vaccine + Durvalumab | Neoantigen DNA Vaccine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With an Immune Response to Neoantigen DNA Vaccines Given Alone or in Combination With Durvalumab as Measured by Interferon-gamma ELISPOT Assay
Description: The ELISpot assay was performed after in vitro culture of patient PBMC with neoantigen peptide for ~12 days. The number of spot-forming T cells, a surrogate for the number of neoantigen-specific T cells, was determined after neoantigen peptide re-stimulation for the duration of the assay (48 hours) and compared to that of control cells that were not re-stimulated with neoantigen during the assay. One-way anova analysis was performed on replicate assessments.
Time Frame: Up to 1 year after completion of treatment (approximately 1 year and 141 days)
Population: 4 participants in the Neoantigen DNA vaccine + Durvalumab arm were not evaluable due to early withdrawal from treatment (2=lack of efficacy, 2=withdrawal by subject). 2 participants in the Neoantigen DNA vaccine arm were not evaluable due to early withdrawal from treatment (1=adverse event, 1=only 5 out of 6 vaccines received).
Measure: Count of Participants; unit: Participants
Arm/Group | Neoantigen DNA Vaccine + Durvalumab | Neoantigen DNA Vaccine
Number analyzed (Participants) | 5 | 7
Participants | 3 | 6

4. Secondary Outcome: Number of Participants With Immune Response to Neoantigen DNA Vaccines Given Alone or in Combination With Durvalumab as Measured by Multiparametric Flow Cytometry - CD4
Description: Multiparametric flow cytometry was performed as a second readout to assess neoantigen-specific T cell reactivity. Markers included CD4, CD8, IFNγ, and a viability marker. After culture, as described above, T cells were stimulated for 6 hours with/without neoantigen and stained with fluorescent antibodies specific for the various markers. Data were analyzed by comparing the percentage IFNγ+ CD4/CD8 cells between neoantigen-stimulated vs unstimulated T cells; a >2-fold increase in percentage positive cells after neoantigen stimulation was considered positive.
Time Frame: Up to 1 year after completion of treatment (approximately 1 year and 141 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Neoantigen DNA Vaccine + Durvalumab | Neoantigen DNA Vaccine
Number analyzed (Participants) | 5 | 7
Participants | 3 | 4

5. Secondary Outcome: Number of Participants With Immune Response to Neoantigen DNA Vaccines Given Alone or in Combination With Durvalumab as Measured by Multiparametric Flow Cytometry - CD8
Description: as for outcome 4
Time Frame: Up to 1 year after completion of treatment (approximately 1 year and 141 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Neoantigen DNA Vaccine + Durvalumab | Neoantigen DNA Vaccine
Number analyzed (Participants) | 5 | 7
Participants | 3 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 90 days after completion of treatment (median follow-up 242 days, full range 132-300 days). All-cause mortality is collected from start of treatment through completion of follow-up (follow-up was a total of 1378 days).
Arm/Group | Neoantigen DNA Vaccine + Durvalumab | Neoantigen DNA Vaccine
All-Cause Mortality (participants affected / at risk) | 1/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 9/9 | 9/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoantigen DNA Vaccine + Durvalumab (N=9) | Neoantigen DNA Vaccine (N=9)
Anemia (Blood and lymphatic system disorders) | 3 | 1
Chest pain-cardiac (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Visual migraine (Eye disorders) | 0 | 1
Abdominal cramps (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2
Ankle edema (General disorders) | 0 | 1
Chills (General disorders) | 2 | 2
Edema limbs (General disorders) | 1 | 1
Fatigue (General disorders) | 3 | 2
Fever (General disorders) | 1 | 2
Flu-like symptoms (General disorders) | 1 | 2
Injection site pain (General disorders) | 9 | 9
Localized edema (General disorders) | 2 | 1
Neck edema (General disorders) | 1 | 0
COVID-19 infection (Infections and infestations) | 1 | 0
Infection from cat bite (Infections and infestations) | 1 | 0
Oral herpes lesions (Infections and infestations) | 0 | 1
Port infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Broken foot (Injury, poisoning and procedural complications) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 3
Neutrophil count decreased (Investigations) | 0 | 2
Weight gain (Investigations) | 0 | 1
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 1 | 2
Neuralgia (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Blanching of fingers on left hand (Skin and subcutaneous tissue disorders) | 0 | 1
Candidal rash (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 1
Nodule on breast (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Bilateral breast fat grafting (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 2 | 3
Lymphedema (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/40/NCT03199040/Prot_SAP_000.pdf